CLINICAL TRIAL: NCT02881684
Title: Weight Reduction by Aspiration Therapy in Asian Patients With Morbid Obesity
Brief Title: Aspiration Therapy in Asian Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Aspire Bariatrics, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Michele Yuen, Specialist in Endocrinology & Metabolism, Honorary Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UW 16-244
Record Dates: First submitted 2016-08-12; First posted 2016-08-29 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Intervention:
  1. Device: Aspiration Therapy (AspireAssist)
     - Subjects randomized to the treatment group will undergo an endoscopic procedure to have the experimental device (i.e. the A-tube) inserted. This will be followed by regular follow up visits and lifestyle therapy matched to the control group. The device will be removed at the end of one year and this group will be observed for one year more to determine if there is any legacy effect.
  2. Behavioral: Lifestyle Therapy Lifestyle therapy is a behavioral, diet and physical activity education program Other Name: Lifestyle Behavioral Therapy
  Interventions: Device: Aspiration Therapy (AspireAssist®); Behavioral: Lifestyle Therapy
- Control (Active Comparator): Intervention:
  (1) Behavioral: Lifestyle Therapy Lifestyle therapy is a behavioral, diet and physical activity education program Other Name: Lifestyle Behavioral Therapy
  - Subjects randomized to the control group will receive lifestyle management matched to the treatment group in the first year. At the end of one year, they will be crossed over to treatment and the A-tube will be inserted. They will then follow up the same follow up schedule of the treatment group during the first year.
  Interventions: Device: Aspiration Therapy (AspireAssist®); Behavioral: Lifestyle Therapy

INTERVENTIONS:
Device: Aspiration Therapy (AspireAssist®) — Use of the AspireAssist device in aspiration therapy
  Other Names: AspireAssist® Aspiration Therapy System
Behavioral: Lifestyle Therapy — Lifestyle therapy is a behavioral, diet and physical activity education program
  Other Names: Lifestyle Behavioral Therapy

SUMMARY:
This research project will provide insight into the efficacy and safety of aspiration therapy in the management of obesity and its comorbidities in the Asian population, and will determine if there is a role for this novel endoscopic device in the treatment algorithm of obesity in the investigators' local regions.

DETAILED DESCRIPTION:
Obesity is a major global health problem and Asians are equally affected. According to the latest Behavioural Risk Factor Survey in 2014, 20.8% of adults in Hong Kong have body mass index (BMI) belonging to the obese category. Obesity is associated with a multitude of medical and psychological comorbidities that could cumulate in increased healthcare costs and impaired quality of life. As such, an effective treatment strategy for obesity is imperative.

Sustainable weight reduction by lifestyle measures alone is often difficult if not impossible. Pharmacotherapy can provide additional weight reduction when used as an adjunct to lifestyle intervention but the efficacy is modest. The most effective method for weight reduction to date is bariatric surgery but this is limited by its invasiveness and irreversibility. The limitations of current obesity treatment has led to an increased interest in endoscopic treatment, which may be more effective than pharmacotherapy and less invasive and more reversible than bariatric surgery.

The AspireAssist® Aspiration Therapy System is a novel endoscopic therapy developed by Aspire Bariatrics Inc. (King of Prussia, United States) for treatment of obesity. The system takes advantage of percutaneous endoscopic gastrostomy (PEG) tube technology to induce weight reduction by aspirating a portion of ingested meals from the stomach. In a pilot study involving 18 Caucasian obese subjects randomly assigned in a 2:1 ratio to aspiration therapy group and lifestyle therapy only group, the weight reduction was 18.6% +/- 2.3% and 5.9% +/- 5.0% respectively. The present study aims to investigate the effectiveness and safety of this device in Asian subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Measured body mass index (BMI) of 27.5-55.0 kg/m2 at time of screening.
2. 21- 65 years of age (inclusive) at time of screening.
3. Failed attempt for a duration equal to 3-months at weight loss by alternative approaches (e.g. supervised or unsupervised diets, exercise, behavioral modification programs)
4. Stable weight (<3% change in self-reported weight) over the previous 3 months at time of screening.
5. Women of childbearing potential who agree to use at least one form of birth control (prescription hormonal contraceptives, diaphragm, intrauterine device (IUD), condoms with or without spermicide, or voluntary abstinence) from time of study enrollment through study exit
6. Willing and able to provide informed consent and comply with the protocol.

Exclusion Criteria:

1. Evidence of an eating disorder or major depression
2. History of gastrointestinal disease or previous gastric surgery that would increase the risk of the AspireAssist® Tube (A-Tube) placement
3. Severe co-existing medical diseases or malignancies
4. Bleeding tendency (low platelet, coagulopathy including being on anti-coagulants)
5. Pregnant/lactating

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Weight reduction by aspiration therapy after 1 year of treatment | 1 year
  Aspiration therapy using the AspireAssist® Aspiration Therapy System (Aspire Bariatrics Inc., King of Prussia, United States) for weight reduction in Asian subjects with obesity over a 12-month treatment period.

SECONDARY OUTCOMES:
Change in blood pressure | 2 years
  mean percent change in systolic and diastolic blood pressures during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in Serum Lipids | 2 years
  mean percent change serum lipids (triglyceride, HDL-cholesterol and LDL-cholesterol concentration) during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in Mean Hemoglobin A1c | 2 years
  change in mean hemoglobin A1C (only subjects with T2 diabetes at baseline) during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in serum leptin | 2 years
  change in mean serum leptin levels during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in serum ghrelin | 2 years
  change in mean serum ghrelin levels during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in serum peptide YY | 2 years
  change in mean serum peptide YY levels during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in serum gastric inhibitory polypeptide | 2 years
  change in mean serum gastric inhibitory polypeptide levels during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in serum glucagon-like peptide 1 | 2 years
  change in mean serum glucagon-like peptide 1 levels during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in serum amylin | 2 years
  change in mean serum amylin levels during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in serum pancreatic polypeptide | 2 years
  change in mean serum pancreatic polypeptide levels during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in serum cholecystokinin | 2 years
  change in mean serum cholecystokinin levels during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in serum insulin | 2 years
  change in mean serum insulin levels during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in serum C-peptide | 2 years
  change in mean serum C-peptide levels during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in serum fibroblast growth factor 19 | 2 years
  change in mean serum fibroblast growth factor 19 levels during treatment (aspiration therapy + lifestyle therapy) period compared to control (lifestyle therapy only) period, and in the AT group compared to the control group
Change in perceived appetite / satiety | 2 years
  Using the control of eating questionnaire
Change in depressive symptoms | 2 years
  Patient Health Questionnaire
Change in anxiety symptoms | 2 years
  State-Trait Anxiety Inventory (STAI)
Change in eating behavior | 2 years
  Eating Disorder Examination (EDE-Q)
Change in psychosocial functioning | 2 years
  Obesity Related Psychological Problem Scale (OP Scale)
Electrolyte disturbances | 2 years
  Number of treatment group subjects with hypokalemia, hypokalemia requiring oral replacement therapy and hypokalemia requiring in-patient care
Micronutrient disturbances | 2 years
  Number of treatment group subjects with iron / vitamin B12 / folate deficiencies, with iron / vitamin B12 / folate deficiencies requiring oral replacement therapy and with iron / vitamin B12 / folate deficiencies requiring in-patient care
Adverse events | 2 years
  The incidence of procedure-related, device-related, and therapy-related adverse events unrelated to electrolyte or micronutrient disturbances will be measured, as well as the incidence of device related, or unrelated, serious adverse events, including unanticipated adverse device effects. Also, the development of adverse eating behaviors will be assessed.
Sustainability of weight reduction (if any) with removal of the A-tube after the treatment period | 1 year
  Mean weight gain during the first year after removal of the A-tube in the AT group

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations for studies involving linear regression. Control Clin Trials. 1998 Dec;19(6):589-601. doi: 10.1016/s0197-2456(98)00037-3. PMID 9875838
- [Background] Ko GT. The cost of obesity in Hong Kong. Obes Rev. 2008 Mar;9 Suppl 1:74-7. doi: 10.1111/j.1467-789X.2007.00442.x. PMID 18307703
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Mond JM, Hay PJ, Rodgers B, Owen C, Beumont PJ. Validity of the Eating Disorder Examination Questionnaire (EDE-Q) in screening for eating disorders in community samples. Behav Res Ther. 2004 May;42(5):551-67. doi: 10.1016/S0005-7967(03)00161-X. PMID 15033501
- [Background] Beumont PJ, Kopec-Schrader EM, Talbot P, Touyz SW. Measuring the specific psychopathology of eating disorder patients. Aust N Z J Psychiatry. 1993 Sep;27(3):506-11. doi: 10.3109/00048679309075810. PMID 8250797
- [Background] Karlsson J, Taft C, Sjostrom L, Torgerson JS, Sullivan M. Psychosocial functioning in the obese before and after weight reduction: construct validity and responsiveness of the Obesity-related Problems scale. Int J Obes Relat Metab Disord. 2003 May;27(5):617-30. doi: 10.1038/sj.ijo.0802272. PMID 12704406
- [Background] van Hout GC, van Oudheusden I, van Heck GL. Psychological profile of the morbidly obese. Obes Surg. 2004 May;14(5):579-88. doi: 10.1381/096089204323093336. PMID 15186623
- [Background] Herpertz S, Kielmann R, Wolf AM, Langkafel M, Senf W, Hebebrand J. Does obesity surgery improve psychosocial functioning? A systematic review. Int J Obes Relat Metab Disord. 2003 Nov;27(11):1300-14. doi: 10.1038/sj.ijo.0802410. PMID 14574339
- [Background] Abiles V, Rodriguez-Ruiz S, Abiles J, Mellado C, Garcia A, Perez de la Cruz A, Fernandez-Santaella MC. Psychological characteristics of morbidly obese candidates for bariatric surgery. Obes Surg. 2010 Feb;20(2):161-7. doi: 10.1007/s11695-008-9726-1. Epub 2008 Oct 29. PMID 18958537
- [Result] Sullivan S, Stein R, Jonnalagadda S, Mullady D, Edmundowicz S. Aspiration therapy leads to weight loss in obese subjects: a pilot study. Gastroenterology. 2013 Dec;145(6):1245-52.e1-5. doi: 10.1053/j.gastro.2013.08.056. Epub 2013 Sep 6. PMID 24012983
- [Result] Pekkarinen T, Kaukua J, Mustajoki P. Long-term weight maintenance after a 17-week weight loss intervention with or without a one-year maintenance program: a randomized controlled trial. J Obes. 2015;2015:651460. doi: 10.1155/2015/651460. Epub 2015 Mar 30. PMID 25918644
- See also: Obesity. Centre for Health Protection, Department of Health, Government of Hong Kong, 2015. — https://www.chp.gov.hk/en/healthtopics/content/25/8802.html